CLINICAL TRIAL: NCT03671447
Title: Enhanced Recovery After Intensive Care (ERIC) - a Multi-Center Stepped Wedge Cluster-Randomized Controlled Trial
Brief Title: Enhanced Recovery After Intensive Care (ERIC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Innovationsausschuss beim Gemeinsamen Bundesausschuss (G-BA), Berlin, Germany (Unknown); Fraunhofer-Institut für Offene Kommunikationssysteme FOKUS, Berlin, Germany (Unknown); BARMER (Other); Klinik Ernst von Bergmann Bad Belzig gGmbH, Bad Belzig, Germany (Unknown); Technische Universität Berlin (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Operative Intensive Care Medicine CCM/CVK, Charite University, Berlin, Germany
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ERIC
Record Dates: First submitted 2018-08-22; First posted 2018-09-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Critical Illness
Keywords: intensive care medicine; critical illness; post intensive care syndrome; e-health; tele-ICU; quality indicators (QIs) in intensive care medicine; German Innovation Fund
MeSH Terms: conditions — Critical Illness; postintensive care syndrome | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Stepped Wedge design with cluster-randomization of sites to 3 sequence groups ("switching groups"). Hereby, sites cross over to the intervention condition sequentially in a random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU usual care (Active Comparator): control condition
  Interventions: Other: ICU Usual Care
- Intervention "ERIC" (Experimental): intervention condition
  Interventions: Behavioral: Tele-ICU

INTERVENTIONS:
Other: ICU Usual Care — The control condition delivered at ICU is usual care.
  Arms: ICU usual care
Behavioral: Tele-ICU — The experimental complex intervention ERIC consists of daily tele-medicine based rounds at ICU. Tele-ICU is implemented after a blended learning program for ICU staff which will be completed prior to the site's crossover.
  Arms: Intervention "ERIC"

SUMMARY:
The primary objective of the multi-center stepped-wedge cluster-randomized controlled trial ERIC is to evaluate the effects of a multi-component telemedicine-based intervention delivered by the ICU on the adherence to quality indicators (QI) in intensive care medicine compared to usual care.

Critically ill patients treated on the interventional condition receive daily tele-medical rounds during their ICU stay.

Further secondary objectives are to demonstrate whether the intervention improves patient outcomes 3 and 6 months post ICU discharge, compared to usual care.

DETAILED DESCRIPTION:
Rationale:

Survivors of critical illness frequently develop long-term mental, cognitive, and/or physical impairments summarized as Post Intensive Care Syndrome (PICS). On the national society level, Germany uses 10 core QIs that are evidence-based to improve treatment quality at ICUs.

Objective:

To investigate whether a tele-medical intervention delivered at ICU improves the adherence to established evidence-based QIs in intensive care medicine compared to the adherence at ICUs delivering usual care.

Study design:

ERIC is a stepped-wedge cluster-randomized controlled quality improvement trial with participating ICUs crossing over from usual care to a multifaceted e-health intervention. After the rollout, all recruiting sites will have implemented the experimental intervention for at least 4 months. Follow-up assessments on the patient-level at month 3 and 6 after ICU discharge (index stay) will be conducted in the outpatient or inpatient setting (dependent on the patient's health status).

Study population:

Critically ill patients covered by statutory health insurance treated at participating ICUs in Berlin and Brandenburg, Germany. It is planned to recruit 1431 study patients within 16 months.

Intervention:

Complex telemedicine-based intervention incorporating the use of e-health technologies (virtual care), supported by blended learning of ICU staff prior to the site's crossover.

Comparison:

Intensive care according to current practice.

Endpoints:

Eight co-primary endpoints will be specified. A primary efficacy endpoint is the adherence to a single QI in intensive care medicine (definition according to Kumpf O. et al., 2017) measured on a daily basis, on a patient-level.

Sedation and delirium management in Frankfurt/Oder before and after implementation of the new form of care ERIC - (SeDelFIN) In this sub-project it should be evaluated how the implementation of the evidence-based standard for delirium, analgesia and pain management changes changed after the introduction of the new form of care. For this purpose, the patient files (which are available in paper form) of all patients who were admitted to the intensive care unit of the Department of Anaesthesiology, Intensive Care Medicine and Pain therapy at the Frankfurt/Oder Clinic (study center) were analyzed by Wilma Klink.

ELIGIBILITY:
Patient Level:

Inclusion Criteria:

* Age ≥ 18 years
* Expected to receive treatment in a medical or surgical ICU connected to the project for more than 24 hours
* Coverage by a German statutory health insurance company
* Written informed consent of patient or legal representative

Exclusion Criteria:

• Age < 18 years

Institutional level:

Inclusion Criteria:

* Located in the Berlin/Brandenburg metropolitan region
* Adherence to general legal obligations to participate in the study funded by the German Innovation Fund and participate in the respective contracts.
* Adherence to cluster-randomization

Exclusion Criteria:

• No intensive care beds available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1463 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-11-17 (Actual)

PRIMARY OUTCOMES:
QI 'Daily multiprofessional and interdisciplinary clinical visits with documentation of daily goals' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Management of sedation, analgesia, and delirium' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Patient-adapted ventilation' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Early weaning from invasive ventilation' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Measures for infection management' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Early enteral nutrition' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Documentation of structured patient and family communications' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level
QI 'Early mobilization' | From enrolment to ICU discharge; Patients assessed for the duration of their ICU stay after enrolment, expected average of 14 days.
  The adherence [fulfilled yes/no] to this intra-hospital QI is daily assessed on a patient-level

SECONDARY OUTCOMES:
All-cause mortality | Up to 6 months following the first study-related ICU admission
  Number of deaths from any cause within 6 months after enrolment including in-hospital mortality will be recorded (using hospital administrative records, electronic medical records, municipal personal records database and the 3- and 6-month follow-up with surrogates).
Mental Health Condition - Depression and Anxiety | 3 and 6 months after ICU discharge
  The patient-reported symptom burden on anxiety and depression will be assessed by the paper-based Patient-Health-Questionnaire PHQ-4 at month 3 and 6. Higher total scores indicate higher impairment.
Mental Health Condition - Post-traumatic Stress | 6 months after ICU discharge
  Patient-reported symptom burden on post-traumatic stress will be assessed by the paper-based questionnaire Impact of Event Scale revised (IES-R) at month 6. Higher total scores indicate greater distress.
Cognition - MiniCog | 3 and 6 months after ICU discharge
  Cognitive functional outcome as assessed by the MiniCog test (2 tests: three-item recall task; clock-drawing task) at month 3 and 6. Higher scores indicate better cognitive functioning.
Cognition - Animal Naming Test | 3 and 6 months after ICU discharge
  Cognitive functional outcome as assessed by the Animal Naming test at month 3 and 6. Higher scores indicate better cognitive functioning.
Physical Function - Timed Up & Go Test | 3 and 6 months after ICU discharge
  Patient's physical function, walking ability and risk of fall as assessed by the Timed Up & Go (TUG) test at month 3 and 6. Higher scores indicate a higher level of impairment.
Physical Function - Hand grip strength test | 3 and 6 months after ICU discharge
  Patient's muscle/ nerve function is assessed by the Hand grip strength (HGS) test (measured with a dynamometer, average strength [in kg] of three trials for the dominant hand) at months 3 and 6.
Health-related quality of life | 3 and 6 months after ICU discharge
  Patient's self-reported health-related quality of life as measured by the EuroQol - 5 Dimensions - 5 Level (EQ-5D-5L) Visual Analogue Scale (VAS) and the EQ-5D-5L descriptive system; the EQ-5D-5L VAS is a thermometer-like rating scale ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Organ dysfunction | 3 and 6 months after ICU discharge
  Number of patients with organ dysfunction as assessed by general practitioner or study personnel/ investigator at month 3 and 6.
Pulmonary Function - Dyspnea | 6 months after ICU discharge
  Self-perceived breathlessness as assessed by the Modified British Medical Research Council (mMRC) Dyspnea Scale at month 6. 5-point Likert scale [range 1 to 5] with a higher score indicating higher impairment.
Outpatient ventilation | Up to 6 months after ICU discharge
  Duration [in days] of mechanical ventilation after discharge from the ICU
Patient-reported Functioning and Disability (WHO Disability Assessment Schedule). | 6 months after ICU discharge
  Patient-reported General Disability Score as measured by the WHO Disability Assessment Schedule (WHODAS 2.0) for activity limitation and participation restriction, 12-item short version, self-administered questionnaire. The raw score is calculated by summing the values for each of the 12 questions. Higher scores indicate greater disability.

OTHER OUTCOMES:
Economic - Length of stay at intensive care unit | Up to 6 months
  Patients will be followed for duration of stay. The total number of days spent in ICU will be assessed (inclusive of index ICU stay).
Economic - Length of hospital stay | Up to 6 months
  Patients will be followed for duration of hospital stay. The total number of days spent in a hospital will be assessed (inclusive of index ICU stay and index hospitalization).
Economic - Return to work | 3 and 6 months after ICU discharge
  Employment status at 3 months and 6 months after hospital discharge (including e.g. return to work, change in duties or change in effectiveness) at 3 and 6 months.
Economic - Cost-effectiveness | 3 and 6 months after ICU discharge
  Health-related costs for standard care and supportive care will be estimated in Euros per patient per months. Data source will be GPs, hospital-electronic health records and health insurance data as well as publicly available data sources from the German reimbursement system.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiolgy and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin
Locations (13):
- Germany (13):
  - Sana Klinikum Lichtenberg, Berlin
  - Department of Anesthesiolgy and Operative Intensive Care Medicine, Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Maria Heimsuchung Caritas Klinik Pankow, Berlin
  - Department of Anesthesiolgy and Operative Intensive Care Medicine CCM/CVK, Charité - Universitätsmedizin Berlin, Berlin
  - Paul Gerhard Diakonie - Evangelisches Waldkrankenhaus Spandau, Berlin
  - Paul Gerhard Diakonie - Evangelisches Krankenhaus Hubertus, Berlin
  - Paul Gerhard Diakonie - Martin-Luther-Krankenhaus, Berlin
  - Klinikum Barnim Werner-Forßmann-Krankenhaus, Eberswalde
  - Klinikum Frankfurt (Oder), Frankfurt (Oder)
  - Ruppiner Kliniken, Neuruppin
  - Ernst von Bergmann Klinikum - Clinic for Anesthesiology and Operative Intensive Care Medicine, Potsdam
  - Ernst von Bergmann Klinikum - Clinic for Emergency and Internal-Intensive Care Medicine, Potsdam

REFERENCES:
- [Background] Kumpf O, Braun JP, Brinkmann A, Bause H, Bellgardt M, Bloos F, Dubb R, Greim C, Kaltwasser A, Marx G, Riessen R, Spies C, Weimann J, Wobker G, Muhl E, Waydhas C. Quality indicators in intensive care medicine for Germany - third edition 2017. Ger Med Sci. 2017 Aug 1;15:Doc10. doi: 10.3205/000251. eCollection 2017. PMID 28794694
- [Background] Kastrup M, Tittmann B, Sawatzki T, Gersch M, Vogt C, Rosenthal M, Rosseau S, Spies C. Transition from in-hospital ventilation to home ventilation: process description and quality indicators. Ger Med Sci. 2017 Dec 19;15:Doc18. doi: 10.3205/000259. eCollection 2017. PMID 29308061
- [Derived] Ribet Buse E, Grunow JJ, Spies CD, Weiss B, Paul N. Health-related quality of life correlates with patient-reported and proxy-reported disability in critical illness survivors: a secondary analysis of the ERIC trial. Crit Care. 2025 Apr 23;29(1):158. doi: 10.1186/s13054-025-05399-3. PMID 40270036
- [Derived] Paul N, Ribet Buse E, Grunow JJ, Schaller SJ, Spies CD, Edel A, Weiss B. Prolonged Mechanical Ventilation in Critically Ill Patients: Six-Month Mortality, Care Pathways, and Quality of Life. Chest. 2025 Jul;168(1):106-118. doi: 10.1016/j.chest.2025.01.018. Epub 2025 Jan 27. PMID 39880302
- [Derived] Paul N, Cittadino J, Krampe H, Denke C, Spies CD, Weiss B. Determinants of Subjective Mental and Functional Health of Critical Illness Survivors: Comparing Pre-ICU and Post-ICU Status. Crit Care Med. 2024 May 1;52(5):704-716. doi: 10.1097/CCM.0000000000006158. Epub 2024 Jan 8. PMID 38189649
- [Derived] Spies CD, Paul N, Adrion C, Berger E, Busse R, Kraufmann B, Marschall U, Rosseau S, Denke C, Krampe H, Dahnert E, Mansmann U, Weiss B; ERIC Study Group. Effectiveness of an intensive care telehealth programme to improve process quality (ERIC): a multicentre stepped wedge cluster randomised controlled trial. Intensive Care Med. 2023 Feb;49(2):191-204. doi: 10.1007/s00134-022-06949-x. Epub 2023 Jan 16. PMID 36645446
- [Derived] Paul N, Cittadino J, Weiss B, Krampe H, Denke C, Spies CD. Subjective Ratings of Mental and Physical Health Correlate With EQ-5D-5L Index Values in Survivors of Critical Illness: A Construct Validity Study. Crit Care Med. 2023 Mar 1;51(3):365-375. doi: 10.1097/CCM.0000000000005742. Epub 2023 Jan 5. PMID 36606801
- [Derived] Adrion C, Weiss B, Paul N, Berger E, Busse R, Marschall U, Caumanns J, Rosseau S, Mansmann U, Spies C; ERIC study group. Enhanced Recovery after Intensive Care (ERIC): study protocol for a German stepped wedge cluster randomised controlled trial to evaluate the effectiveness of a critical care telehealth program on process quality and functional outcomes. BMJ Open. 2020 Sep 25;10(9):e036096. doi: 10.1136/bmjopen-2019-036096. PMID 32978185
- See also: Quality indicators in intensive care medicine for Germany - third edition 2017 — https://www.egms.de/static/en/journals/gms/2017-15/000251.shtml
- See also: Funding source body of study — https://www.g-ba.de/english/